CLINICAL TRIAL: NCT05597319
Title: Enhanced Recovery After Surgery: Compliance to the Program in Liver Surgery and Factors Associated With Drop-out
Brief Title: ERAS in Liver Surgery
Acronym: ERASliver
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: ERASliver
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: ERAS
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS-in: Patients who completed ERAS program
  Interventions: Procedure: Liver resection
- ERAS-out: Patients who dropped-out from ERAS program
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Liver resection, different kind of according to pathology

SUMMARY:
Enhanced Recovery After Surgery (ERAS) Program (EP) is widely applied to obtain a reduction in post-operative length of hospital stay and a faster restoration of pre-operative patient conditions. However, in Western countries, adherence to EP in liver surgery is still difficult to achieve due to deep-rooted traditional practices. In our Institute, since 2019, EP has been applied pursuing 18/23 items identified by 2016 guidelines. At all consecutive patients who underwent elective liver surgery in our Institution, EP was proposed and their adherence to ERAS items was measured before, during and after surgery. Data were retrospectively collected and analysed, particularly focusing on EP items. Primary outcome was compliance to EP, defined as at least 80% of accomplished items per patient. Secondary outcome was adherence to each ERAS item, while tertiary outcome was detecting the variables associated with program drop out.

ELIGIBILITY:
Inclusion Criteria:

* patients candidates to surgery for benign or malignant liver disease
* liver resection with curative intent

Exclusion Criteria:

* refusal to participate at the EP
* incapability to acquire informed consent
* cognitive impairment that can prejudice the patient comprehension of the EP
* liver surgery with palliative or diagnostic intent or non-resective liver surgery
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 126 patients were consecutively enrolled from January 2019 to July 2021
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Compliance to ERAS program | 32 months
  Compliance to ERAS program was defined as at least 80% of accomplished items per patient

SECONDARY OUTCOMES:
Compliance to ERAS items | 32 months
  Compliance to each ERAS item singularly
Drop-out factors | 32 months
  Determining factors associated with ERAS program drop-out

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Gerardo, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No